CLINICAL TRIAL: NCT05013762
Title: Fast Training Promotes Recovery of Arm Movements Post-stroke Via Cerebellar-mediated Anticipatory Feedforward Control
Brief Title: Fast Arm Motor Skill Training
Acronym: FAST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: Casa Colina Hospital and Centers for Healthcare (Other)
Responsible Party: Principal Investigator, Carolee Winstein, Professor, Biokinesiology and Physical Therapy, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HS-CG-20-00023
Record Dates: First submitted 2021-07-02; First posted 2021-08-19 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Cerebrovascular Stroke
Keywords: Stroke; Physical therapy; neurorehabilitation; motor function; neuroplasticity; neuroimaging; MRI; TDI; Hemiparesis; occupational therapy; patient focused; motor learning; motor control; skill acquisition; skill training; motor recovery; task-oriented training; task-specific training; arm function; upper extremity; arm therapy; physical rehabilitation; arm rehabilitation
MeSH Terms: conditions — Stroke; Paresis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Assessments will be done by a blinded and standardized clinical researcher
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Speed-biased complex motor skill training (Active Comparator): Participants will perform 400 complex movements per day over 4 days over a one-week period. The task requires participants to navigate their hand through a "track" projected on the surface of a table with a width of 5cm. Participants receive adaptive score based on their movement time. .
  Interventions: Behavioral: Fast intervention
- Accuracy-biased complex motor skill training (Other): The accuracy-biased group receives a dose equivalent intervention with a emphasize on accuracy. The width of the track projected on the table is narrower (less than 2cm) and the adaptive score received are based on their accuracy to say within the boundary of the track.
  Interventions: Behavioral: Active Monitoring

INTERVENTIONS:
Behavioral: Fast intervention — This intervention is based on recent body of evidence that high-speed movements during training are effective at improving arm movements in individuals with chronic stroke.Participants will be rewarded for movements performed within a short amount of time.
  Arms: Speed-biased complex motor skill training
Behavioral: Active Monitoring — This is an observation-only group. The training received in this group will be dose equivalent to the active group.
  Arms: Accuracy-biased complex motor skill training

SUMMARY:
Every year, almost 800,000 people experience a stroke in the United States, which lead to upper-limb impairments, making recovery of motor function a priority in stroke rehabilitation. 1) The primary objective of this study is to determine whether fast arm movement training on a tracking task ("Speed-training"), in chronic stroke survivors with mild to moderate paresis, will generalize to improve arm function better than dose-equivalent accuracy training on the same task. 2) study the effect of intensive arm training on the recovery of anticipatory feedforward control. 3) Determine the involvement of cerebellar-cortical circuits in the recovery of arm movements due to speed training.

DETAILED DESCRIPTION:
About 65% of stroke survivors experience long-term limitations in upper extremity (UE) functions. In particular, limitations in arm reaching movements are prominent and correlate strongly with patients' impairment levels. Because activities of daily living often involve the UEs, retraining reach and grasp skills is critical for return to a full quality-of-life. Yet, the training parameters required for effective rehabilitation of UE function are not known. Recent evidence suggests that high-speed movements during training are effective at improving arm movements in individuals with chronic stroke. Hence, fast movements generating large errors, would promote the restoration of the feedforward controllers and therefore improves arm movements and UE functions in individuals with chronic stroke. Because the cerebellum is involved in learning feedforward controllers from motor errors, the improvements would be proportional to the integrity of the cerebellar-cortical networks.

A double-blind quasi-randomized controlled study will be carried out in chronic post-stroke survivors. Participants will be assigned to either the speed-bias training group or a dose equivalent accuracy-bias training group (control) and will receive 4 days of training over a 1week period by a trained Occupational or physical therapist. Behavioral, EMG, and MRI data will be acquired within two weeks before, 3 days post, and one month after intervention.

ELIGIBILITY:
Inclusion Criteria:

* At least 6 months following an ischemic supratentorial stroke
* At least 21 years of age
* Exhibit residual capability to move the paretic UE (Upper Extremity Fugl- Meyer motor score >20/66)
* Able to follow a 2-step command (8th item on the MMSE test)
* Able to perform an unassisted arm reach movement of 25 cm ahead of the body within 5 seconds with trunk restraint
* Exhibit no greater than mild/moderate spasticity as assessed with a Modified Ashworth Score < 3

Exclusion Criteria:

* any neurologic diagnoses other than stroke
* peripheral movement restrictions, such as neuropathy
* orthopedic disorders affecting the paretic UE
* severe pain or sensory/proprioceptive impairment in the more affected UE
* visual neglect (more than 4% of lines left uncrossed on Albert's test).
* had a stroke directly affecting the cerebellum
* any contra-indications to MRI scanning
* mostly resolved impairments with an Upper Extremity Fugl- Meyer motor score >58/66

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2021-06-15 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-11-27 (Actual)

PRIMARY OUTCOMES:
Change in arm reaching movement time. | Change from baseline to 3 days post-intervention
  Average movement time for 30 planar reaching movements to target arrayed on a planar workspace.
Change in movement smoothness | Change from baseline to 3 days post-intervention
  Average movement smoothness for 30 planar reaching movements to target arrayed on a planar workspace. Smoothness is computed by number of peaks in hand tangential velocity profiles of arm-reaching movements.
Change in speed Accuracy Trade-off | Change from baseline to 3 days post-intervention
  The investigators will compute the "Fitts" slope between "index of difficulty" of reaching movements and movement time, for targets at 3 distances and of 4 diameters.
Change in arm reaching movement time. | Change from baseline to 1 month post-intervention
  Average movement time for 30 planar reaching movements to target arrayed on a planar workspace.
Change in movement smoothness | Change from baseline to 1 month post-intervention
  Average movement smoothness for 30 planar reaching movements to target arrayed on a planar workspace. Smoothness is computed by number of peaks in hand tangential velocity profiles of arm-reaching movements.
Change in speed Accuracy Trade-off | Change from baseline to 1 month post-intervention
  The investigators will compute the "Fitts" slope between "index of difficulty" of reaching movements and movement time, for targets at 3 distances and of 4 diameters.

SECONDARY OUTCOMES:
Change in Action Research Arm Test (ARAT) | Change from baseline to 3 days post-intervention
  The ARAT assess specific changes in limb function among individuals who sustained a stroke.
Change in Upper Extremity Fugl-Meyer (UEFM) | Change from baseline to 3 days post-intervention
  A test of motor function for the arm that is most affected by the stroke.
Change in Box and Block test score (BBT) | Change from baseline to 3 days post-intervention
  The Box and Block Test (BBT) measures unilateral gross manual dexterity.
Change in Action Research Arm Test (ARAT) | Change from baseline to 1 month post-intervention
  The ARAT assess specific changes in limb function among individuals who sustained a stroke.
Change in Upper Extremity Fugl-Meyer (UEFM) | Change from baseline to 1 month post-intervention
  A test of motor function for the arm that is most affected by the stroke.
Change in Box and Block test score (BBT) | Change from baseline to 1 month post-intervention
  The Box and Block Test (BBT) measures unilateral gross manual dexterity.

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Schweighofer, PhD, Principal Investigator — University of Southern California
Locations (1):
- Casa Colina Hospital and Centers for Healthcare, Pomona, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lang CE, Strube MJ, Bland MD, Waddell KJ, Cherry-Allen KM, Nudo RJ, Dromerick AW, Birkenmeier RL. Dose response of task-specific upper limb training in people at least 6 months poststroke: A phase II, single-blind, randomized, controlled trial. Ann Neurol. 2016 Sep;80(3):342-54. doi: 10.1002/ana.24734. Epub 2016 Aug 16. PMID 27447365
- [Background] Winstein C, Kim B, Kim S, Martinez C, Schweighofer N. Dosage Matters. Stroke. 2019 Jul;50(7):1831-1837. doi: 10.1161/STROKEAHA.118.023603. Epub 2019 Jun 5. PMID 31164067
- [Background] Park H, Kim S, Winstein CJ, Gordon J, Schweighofer N. Short-Duration and Intensive Training Improves Long-Term Reaching Performance in Individuals With Chronic Stroke. Neurorehabil Neural Repair. 2016 Jul;30(6):551-61. doi: 10.1177/1545968315606990. Epub 2015 Sep 24. PMID 26405046
- [Background] Kantak S, McGrath R, Zahedi N, Luchmee D. Behavioral and neurophysiological mechanisms underlying motor skill learning in patients with post-stroke hemiparesis. Clin Neurophysiol. 2018 Jan;129(1):1-12. doi: 10.1016/j.clinph.2017.10.010. Epub 2017 Nov 8. PMID 29127826
- [Background] Pantano P, Baron JC, Samson Y, Bousser MG, Derouesne C, Comar D. Crossed cerebellar diaschisis. Further studies. Brain. 1986 Aug;109 ( Pt 4):677-94. doi: 10.1093/brain/109.4.677. PMID 3488093
- [Background] Kawato M, Gomi H. A computational model of four regions of the cerebellum based on feedback-error learning. Biol Cybern. 1992;68(2):95-103. doi: 10.1007/BF00201431. PMID 1486143
- [Background] Gribble PL, Ostry DJ. Compensation for interaction torques during single- and multijoint limb movement. J Neurophysiol. 1999 Nov;82(5):2310-26. doi: 10.1152/jn.1999.82.5.2310. PMID 10561408
- [Background] Maeda RS, Cluff T, Gribble PL, Pruszynski JA. Feedforward and Feedback Control Share an Internal Model of the Arm's Dynamics. J Neurosci. 2018 Dec 5;38(49):10505-10514. doi: 10.1523/JNEUROSCI.1709-18.2018. Epub 2018 Oct 24. PMID 30355628
- [Derived] Darmon Y, Kantak S, Cone H, Fullmer N, Ouellette D, Winstein C, Rosario ER, Schweighofer N. Speed-Biased Training Temporarily Improves Motor Performance of the Paretic Arm Compared to Accuracy-Biased Training in Chronic Stroke Survivors: The Phase 1 FAST Randomized Clinical Trial. Neurorehabil Neural Repair. 2025 Jul;39(7):542-554. doi: 10.1177/15459683251331582. Epub 2025 May 10. PMID 40346836